CLINICAL TRIAL: NCT03586050
Title: A Study to Evaluate the Safety and Effectiveness of Microwave Ablation in Patients With Hepatocellular Carcinoma in Korea
Brief Title: Study to Evaluate the Safety and Effectiveness of Microwave Ablation in Patients With Hepatocellular Carcinoma in Korea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU_2017_01
Record Dates: First submitted 2018-02-08; First posted 2018-07-13 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-06

CONDITIONS: Carcinoma, Hepatocellular; Hepatocellular Carcinoma; Hepatocellular Cancer; Cancer, Hepatocellular
Keywords: Hepatocellular Carcinoma; liver cancer; cancer; liver
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microwave Ablation (Experimental): All patients will receive microwave ablation using the NeuWave Microwave Ablation System and Accessories
  Interventions: Device: Microwave ablation

INTERVENTIONS:
Device: Microwave ablation — All patients will receive microwave ablation using the NeuWave Microwave Ablation System and Accessories

SUMMARY:
This is a single arm, non-randomized, single center study to evaluate ablation, oncologic outcomes and safety in the treatment of hepatocellular carcinoma.

DETAILED DESCRIPTION:
This prospective, single-arm single center study will provide clinical data for the Neuwave Medical Microwave Ablation System and accessories.

Individuals who undergo microwave ablation of liver tumors who meet study entry criteria, will be enrolled.

The enrollment for the study will continue until 30 eligible subjects complete the 3-month visit after ablation for the primary effectiveness and safety analysis.

The subjects will be followed for approximately up to 36 months after the ablation procedure for safety, oncologic and ablation outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed hepatocellular carcinoma, tumor size of more than 2 cm and up to 5cm, single location, Barcelona Clinic Liver Cancer (BCLC) Stage A based on imaging and biopsy confirmation
2. Primary hepatocellular carcinoma or recurrent hepatocellular carcinoma which was previously treated with ablation or surgical resection only;
3. Scheduled for microwave ablation of the liver;
4. Performance status 0-1 (Eastern Cooperative Oncology Group classification);
5. Functional hepatic reserve based on the Child-Pugh score (Class A or B);
6. American Society of Anesthesiologists (ASA) score < 3;
7. Given voluntary, written informed consent to participate in this study and has authorized the transfer of his/her information to the Sponsor, and willing to comply with study-related evaluation and treatment schedule;
8. At least 19 years of age

Exclusion Criteria:

1. Active bacterial infection or fungal infection;
2. Systemic administration of steroids, including herbal supplements that contain steroids, within 30 days prior to the study procedure;
3. Chemotherapy or radiation therapy for hepatocellular carcinoma may not be performed for 30 days prior to the study procedure;
4. Subject with implantable pacemakers or other electronic implants;
5. Planned/ scheduled liver surgery.
6. Subject with a platelet count of less than 20,000/mm3;
7. Subject with an INR greater than 1.5;
8. Subject with renal failure on renal dialysis;
9. Scheduled concurrent procedure other than microwave ablation in the liver;
10. Pregnant or lactating;
11. Physical or psychological condition which would impair study participation;
12. Participation in any other clinical study concurrently or within the last 3 months;
13. The subject is judged unsuitable for study participation by the Investigator for any other reason;
14. Unable or unwilling to attend follow-up visits and examinations.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2023-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyunchul Rhim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from 04Dec2017 through 21May2020.
Groups:
- Microwave Ablation: Participants underwent microwave ablation using the NEUWAVE Certus 140 2.45 Gigahertz (GHz) Ablation System of liver tumors (Hepatocellular Carcinoma [HCC]) at a single visit, in accordance with their institution's standard-of-care (SOC) for ablation. The treating physician determined the ablation time and power used on a case-by-case basis.
Period: Overall Study
Arm/Group | Microwave Ablation
Started | 33
Full Analysis Set (FAS) | 30
Completed | 28
Not Completed | 5
Not completed — Death | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age of participant at the time of informed consent
  Years | 63.6 (8.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 33
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Maximum Tumor Dimension [Mean (Standard Deviation); unit: Centimeters (cm)] | 2.49 (0.578)
Liver Segment [Count of Participants; unit: Participants] — Location of the tumor in the liver (multiple could be selected)
  Participants
    Segment 3 | 3
    Segment 4 | 6
    Segment 5 | 5
    Segment 6 | 5
    Segment 7 | 6
    Segment 8 | 14
Tumor Depth [Count of Participants; unit: Participants]
  Superficial | 17
  Deep | 9
  Dome | 7
Major Vessel/Duct Assessment [Count of Participants; unit: Participants] — Location of the tumor/ablation in relation to a major vessel/duct
  Participants
    Near Major Vessel/Duct | 14
    No Major Vessel/Duct Near Ablation | 19
BCLC (Barcelona Clinic Liver Cancer) Staging [Count of Participants; unit: Participants] — All participants were confirmed to have BCLC staging of Stage A within 5 weeks prior to the day of ablation based on imaging and biopsy confirmation in accordance with their institution Standard of Care (SOC). The BCLC staging system is validated and widely accepted as it offers the most prognostic information (that is, includes information on tumor size/burden, liver function, and participant's Eastern Cooperative Oncology Group [ECOG] performance status). BCLC stages include 0, A, B, C and D.
  Participants
    0 (Very early stage disease; Child-Pugh score of A, ECOG 0-1, single tumor < 2cm) | 0
    A (Early stage disease; Child-Pugh score of A/B, ECOG 0-1, single or 2-3 tumors < 3cm) | 33
    B (Intermediate stage disease; Child-Pugh score of A/B, ECOG 0-1, multinodular tumors) | 0
    C (Advanced stage disease; Child-Pugh score of A/B, ECOG 0-2, portal vein invasion) | 0
    D (Terminal disease; Child-Pugh score C, ECOG>2, metastasized tumors to lymph nodes or other organs) | 0
Child-Pugh Score [Count of Participants; unit: Participants] — All participants were confirmed to have functional hepatic reserve based on the Child-Pugh score (Class A or Class B) within 5 weeks prior to the day of ablation. Child-Pugh Scores assess the prognosis of liver disease. Five clinical features are assessed and assigned 1-3 points depending on severity (1 being none, 2 being mild, and 3 being severe): encephalopathy, presence of ascites, bilirubin blood level, albumin blood level, and prothrombin time prolongation. Classes A, B, and C are based on the total number of points.
  Participants
    Class A (mild liver disease; 5-6 points) | 30
    Class B (moderately severe liver disease; 7-9 points) | 3
    Class C (severe liver disease; 10-15 points) | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whose Ablation Resulted in Technical Success
Description: Number of participants whose ablation resulted in technical success were reported. Technical success was defined as complete tumor ablation with adequate or insufficient margin, based on contrast-enhanced Magnetic resonance imaging (MRI) and Computed scans immediately following the ablation procedure on Day 0 evaluated by the independent reviewer and principle investigator (PI) based on the response to the question "Confirm outcome of ablation".
Time Frame: Post ablation procedure (Day 0) up to 4 days
Population: FAS included all participants in whom the microwave ablation procedure was completed and who provided information on ablation margins for evaluation of technical success and technique efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
Participants
  PI Assessment | 30
  Independent Reviewer Assessment | 30

2. Secondary Outcome: Number of Participants Whose Ablation Resulted in Primary Technique Efficacy
Description: Number of participants whose ablation resulted in primary technique efficacy were reported. Primary technique efficacy was defined as a complete tumor ablation with adequate or insufficient ablation margin, based on contrast-enhanced MRI and CT scans follow-up at 1 month after the ablation procedure, evaluated by the independent reviewer and PI based on the response to the question "Confirm outcome of ablation". The primary technique efficacy was achieved if responses were either "Complete tumor ablation with adequate margin" or "Complete tumor ablation with insufficient margin".
Time Frame: At 1 month after the ablation procedure on Day 0
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
Participants
  PI Assessment | 30
  Independent Reviewer Assessment | 30

3. Secondary Outcome: Percentage of Participants With Local Tumor Progression (LTP)
Description: Percentage of participants with LTP were reported. The first LTP rate was defined as one minus primary efficacy rate. Primary efficacy rate was defined as percentage of participants with target tumors successfully eradicated following the ablation procedure and measured at each follow-up visit post-ablation. Primary efficacy was achieved when any target tumor had been successfully ablated at the Visit 2 ablation (Technical success achieved) and had no evidence of local tumor progression (LTP) based on the independent reviewer's assessment and PI assessment.
Time Frame: At 1, 3, 6, 9, 12, 18, 24, 30 and 36 months post ablation on Day 0
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
percentage of participants
  PI Assessment: 1 Month post ablation | 0.0
  PI Assessment: 3 Months post ablation | 0.0
  PI Assessment: 6 Months post ablation | 0.0
  PI Assessment: 9 Months post ablation | 0.0
  PI Assessment: 12 Months post ablation | 0.0
  PI Assessment: 18 Months post ablation | 0.0
  PI Assessment: 24 Months post ablation | 3.6
  PI Assessment: 30 Months post ablation | 7.6
  PI Assessment: 36 Months post ablation | 7.6
  Independent Reviewer: 1 Month post ablation | 0.0
  Independent Reviewer: 3 Months post ablation | 0.0
  Independent Reviewer: 6 Months post ablation | 0.0
  Independent Reviewer: 9 Months post ablation | 0.0
  Independent Reviewer: 12 Months post ablation | 0.0
  Independent Reviewer: 18 Months post ablation | 0.0
  Independent Reviewer: 24 Months post ablation | 3.6
  Independent Reviewer: 30 Months post ablation | 7.3
  Independent Reviewer: 36 Months post ablation | 7.3

4. Secondary Outcome: Percentage of Participants With Primary Efficacy
Description: Percentage of participants with primary efficacy based on the independent reviewer and PI assessment were reported. Primary efficacy rate was defined as percentage of participants with target tumors successfully eradicated following the ablation procedure and measured at each follow-up visit post-ablation. Primary efficacy was achieved when any target tumor had been successfully ablated at the Visit 2 ablation (Technical success achieved) and had no evidence of LTP based on the independent reviewer's assessment and PI assessment.
Time Frame: At 1, 3, 6, 9, 12, 18, 24, 30 and 36 months post ablation on Day 0
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
percentage of participants
  PI Assessment: 1 Month post ablation | 100.0
  PI Assessment: 3 Months post ablation | 100.0
  PI Assessment: 6 Months post ablation | 100.0
  PI Assessment: 9 Months post ablation | 100.0
  PI Assessment: 12 Months post ablation | 100.0
  PI Assessment: 18 Months post ablation | 100.0
  PI Assessment: 24 Months post ablation | 96.4
  PI Assessment: 30 Months post ablation | 92.4
  PI Assessment: 36 Months post ablation | 92.4
  Independent Reviewer: 1 Month post ablation | 100.0
  Independent Reviewer: 3 Months post ablation | 100.0
  Independent Reviewer: 6 Months post ablation | 100.0
  Independent Reviewer: 9 Months post ablation | 100.0
  Independent Reviewer: 12 Months post ablation | 100.0
  Independent Reviewer: 18 Months post ablation | 100.0
  Independent Reviewer: 24 Months post ablation | 96.4
  Independent Reviewer: 30 Months post ablation | 92.7
  Independent Reviewer: 36 Months post ablation | 92.7

5. Secondary Outcome: Percentage of Participants With Secondary Efficacy
Description: Percentage of participants with secondary efficacy based on the independent reviewer and PI assessment were reported. Secondary efficacy rate was defined as percentage of participants with target tumors that had undergone successful repeat ablation following identification of local tumor progression.
Time Frame: From time of first ablation (Day 0) up to 36 months
Population: FAS included all participants in whom the microwave ablation procedure was completed and who provided information on ablation margins for evaluation of technical success and technique efficacy. Data for this outcome measure was not collected and analyzed as no participant had undergone repeat ablations.
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 0

6. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: PFS rate was defined as the percentage of participants with PFS. PFS was defined as the time from the first ablation until LTP (first LTP rate was defined as one minus primary efficacy rate), any identification of a new (nontarget) lesion/tumor during follow-up, or death due to any cause (whichever occurs first). PFS rate based on independent reviewer's assessment and PI assessment was reported.
Time Frame: At 36 months after the ablation procedure on Day 0
Population: FAS included all participants in whom the microwave ablation procedure was completed and who provided information on ablation margins for evaluation of technical success and technique efficacy. Here "N" (number of participants analyzed) signifies the number of participants that were evaluable for this outcome measure and "n"(number analyzed) signifies the number of participants analyzed for specified categories.
Measure: Number; unit: Percentage of participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 18
Percentage of participants
  PI Assessment: number analyzed (Participants) | 17
  PI Assessment | 40.8
  Independent Reviewer Assessment | 38.5

7. Secondary Outcome: Overall Survival (OS) Rate
Description: OS rate was defined as the percentage of participants with OS. OS was defined as the time from the first ablation until death due to any cause.
Time Frame: At 36 months after the ablation procedure on Day 0
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
percentage of participants | 90.0

8. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) Within 3 Months Post Ablation
Description: Percentage of participants with AEs within 3 months post ablation were reported. An AE was an untoward medical occurrence (sign, symptom or disease) in a participant, and which did not necessarily have a causal relationship with the study medical device.
Time Frame: From time of first ablation (Day 0) up to 3 months post ablation
Population: Safety analysis set (SAF) included all participants in whom the microwave ablation procedure was attempted, that is, started and regardless of whether it got completed as planned or not.
Measure: Number; unit: percentage of participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 33
percentage of participants | 66.7

9. Secondary Outcome: Percentage of Participants With Adverse Events Within 36 Months Post Ablation
Description: Percentage of participants with AEs within 36 months post ablation were reported. An AE was an untoward medical occurrence (sign, symptom or disease) in a participant, and which did not necessarily have a causal relationship with the study medical device.
Time Frame: From time of first ablation (Day 0) up to 36 months post ablation
Population: SAF included all participants in whom the microwave ablation procedure was attempted, that is, started and regardless of whether it got completed as planned or not.
Measure: Number; unit: percentage of participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 33
percentage of participants | 66.7

10. Secondary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Pain Score
Description: Change from baseline in VAS pain scores were reported. VAS pain score was a self-reported pain score on a 100 millimeter (mm) scale which ranged from ranged from 0 mm (no pain) to 100 mm (severe pain). Higher score indicated severe pain. Baseline was defined as the last non-missing measurement taken prior to date of first microwave ablation (including unscheduled assessments) or on the date of first microwave ablation but prior to the time of first probe placement.
Time Frame: Baseline (Pre-Ablation), Day 0 (post ablation), Months 1, 3, 6, 9, 12, 18, 24, 30 and 36 (post ablation on Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
Score on a scale
  Post ablation (Day 0) | 0.32 (0.258)
  1 Month post ablation | -0.01 (0.194)
  3 Months post ablation | 0.00 (0.204)
  6 Months post ablation | 0.02 (0.214)
  9 Months post ablation | 0.01 (0.211)
  12 Months post ablation | -0.03 (0.176)
  18 Months post ablation | -0.06 (0.145)
  24 Months post ablation | -0.06 (0.148)
  30 Months post ablation | -0.06 (0.121)
  36 Months post ablation | -0.06 (0.180)

11. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30 Scale Score
Description: Change from baseline in EORTC QLQ-C30 scale score were reported. EORTC QLQ-C30 contains 30 questions for assessing overall health in cancer patients. The questions reflect how patients felt during the past week and are scored 1-4 (1=not at all, 2=a little, 3=quite a bit, 4=very much) except for the last two questions, which are scored on a 7-point Likert Scale from 1-7 (1=very poor to 7=excellent). All the questions were transformed to a 0-100 scale and summed for an overall quality of life score, with a high score representing higher quality of life. Baseline: last non-missing measurement prior to date of first microwave ablation or on date of first microwave ablation but prior to time of first probe placement.
Time Frame: Baseline (Pre-Ablation), Months 1, 3, 6, 9, 12, 18, 24, 30 and 36 (post ablation on Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
score on a scale
  1 Month post ablation | 1.23 (11.415)
  3 Months post ablation | -0.05 (11.120)
  6 Months post ablation | -0.42 (14.147)
  9 Months post ablation | 0.74 (14.427)
  12 Months post ablation | 2.23 (9.526)
  18 Months post ablation | 3.38 (13.608)
  24 Months post ablation | 1.59 (15.425)
  30 Months post ablation | 4.01 (11.652)
  36 Months post ablation | 2.47 (13.793)

12. Secondary Outcome: Change From Baseline in EORTC QLQ HCC 18 Scale Score
Description: Change from baseline in EORTC QLQ HCC 18 scale score were reported. EORTC 18-item hepatocellular cancer health-related quality of life questionnaire (QLQ-HCC18) was an 18-multi-item scales which were grouped into 8 symptom scales such as fatigue, body image, jaundice, nutrition, pain, fever, abdominal swelling and sex life. All scales were grouped and converted to scores of 0 to 100 according to the scoring manual; a higher score represented a more severe symptom or problem. Baseline was defined as the last non-missing measurement taken prior to date of first microwave ablation (including unscheduled assessments) or on the date of first microwave ablation but prior to the time of first probe placement.
Time Frame: Baseline (Pre-Ablation), Months 1, 3, 6, 9, 12, 18, 24, 30 and 36 (post ablation on Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
score on a scale
  1 Month post ablation | 1.58 (10.397)
  3 Months post ablation | 1.85 (9.663)
  6 Months post ablation | 0.69 (9.575)
  9 Months post ablation | 1.36 (12.508)
  12 Months post ablation | 1.11 (8.902)
  18 Months post ablation | 3.24 (13.080)
  24 Months post ablation | 0.41 (13.593)
  30 Months post ablation | -1.57 (10.948)
  36 Months post ablation | -4.33 (14.320)

13. Secondary Outcome: Health Economics: Complete Procedure Time
Description: Complete procedure time was defined as the time between the first probe placement and the last probe removal.
Time Frame: Day 0 (On day of ablation treatment)
Population: as for outcome 1
Measure: Median (Full Range); unit: minutes
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
minutes | 19 [4.0 to 46.0]

14. Secondary Outcome: Health Economics: Total Ablation Duration
Description: Total ablation duration were reported.
Time Frame: Day 0 (On the day of ablation treatment)
Population: as for outcome 1
Measure: Median (Full Range); unit: minutes
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
minutes | 7.76 [4.0 to 16.2]

15. Secondary Outcome: Health Economics: Median Number of Ablations
Description: The median number of ablations was reported.
Time Frame: Day 0 (On the day of ablation treatment)
Population: as for outcome 1
Measure: Median (Full Range); unit: ablations
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
ablations | 2 [1 to 5]

16. Secondary Outcome: Health Economics: Length of Hospital Stay
Description: Length of hospital stay were reported. Length of hospital stay was defined as the time from procedure completion to hospital discharge.
Time Frame: Day 0 (On day of ablation treatment) up to 30 days (1-month post ablation visit)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
days | 2 [2 to 22]

17. Secondary Outcome: Health Economics: Percentage of Participants With Single and Multi Probes Usage
Description: Percentage of participants with single and multiple probes usage were reported. PR and LK probes were used at least once.
Time Frame: Day 0 (On the day of ablation treatment)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Microwave Ablation
Number analyzed (Participants) | 30
percentage of participants
  Single probe | 3.3
  Multi probe | 96.7

ADVERSE EVENTS:
Time Frame: From time of first ablation (Day 0) up to 36 months post ablation
Description: SAF included all participants in whom the microwave ablation procedure was attempted, that is started and regardless of whether it got completed as planned or not.
Arm/Group | Microwave Ablation
All-Cause Mortality (participants affected / at risk) | 3/33
Serious Adverse Events (participants affected / at risk) | 7/33
Other Adverse Events (participants affected / at risk) | 22/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microwave Ablation (N=33)
Pyrexia (General disorders) | 1 (1)
Extra nodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microwave Ablation (N=33)
Nausea (Gastrointestinal disorders) | 3 (3)
Pyrexia (General disorders) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 15 (15)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hepatic infarction (Hepatobiliary disorders) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Blood pressure decreased (Investigations) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT03586050/Prot_SAP_000.pdf